CLINICAL TRIAL: NCT06579716
Title: Whole-Body Vibration Versus Kineso Tape on Nerve Conduction in Patient With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamis Samir Ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005322
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional balance exercise + Resistance exercise + Whole-body vibration (Experimental): It consisted of 30 participants diagnosed as having diabetic peripheral neuropathy. Each received traditional balance exercise, resistance exercise, and whole-body vibration, for 6 weeks.
  Interventions: Other: Traditional balance exercise; Other: Resistance exercise; Other: Whole-body vibration (WBV)
- Traditional balance exercise + Resistance exercise + Kineso tape (Experimental): It consisted of 30 participants diagnosed as having diabetic peripheral neuropathy. Each received traditional balance exercise, resistance exercise, and kineso tape, for 6 weeks.
  Interventions: Other: Traditional balance exercise; Other: Resistance exercise; Other: Kineso tape

INTERVENTIONS:
Other: Traditional balance exercise — All patients in both group received a traditional balance exercise program, 3 sessions per week, for 6 weeks. Each session of exercise comprised 10 min of warm-up, 40min of balance exercise, and 5min of cool down. Warm-up included treadmill walking. Balance exercise comprised two sets of sit to stand, one leg stance, tandem stance and 30 squats. The first set of exercises was performed on a stable surface, whereas the second set of exercises was performed on an unstable surface by using Thera band stability trainer. Each set of each exercise was performed for 3 min, with 1-2 min of rest in between the exercises. Cool-down included deep breathing, abdominal breathing, and mild stretching.
Other: Resistance exercise — All patients in both group received a resistance exercise program, 3 sessions per week, for 6 weeks. Each patient was seated in sitting position and the weight sandbags was applied at the dorsum of the foot. The resistance was set to be around 40%-60% of the 1RM. The patient performed the exercise for 3 bouts, every bout 10 repetitions. The one repetition maximum (1RM) was established prior to the training period using the following equation: 1 RM = Weight (kg) X (1 + {0.033 X number of repetitions)}.
Other: Whole-body vibration (WBV) — Patients were asked to stand barefoot on the vibratory platform with an even distribution of weight on both feet and familiarized with WBV at a lesser frequency and amplitude. Then, they were asked to bend their knee 30º to the vertical; thereafter, to obtain a greater muscular response, WBV training was performed at a frequency of 30 Hz and an amplitude of 2mm. The exercise comprised five bouts of a 30-sec vibration with a 1-min elapse between the bouts.
  Arms: Traditional balance exercise + Resistance exercise + Whole-body vibration
Other: Kineso tape — Kineso tape was applied to dorsiflexors 24 hours a day and was replaced every 5 days for patients who were taped in accordance with Kenzo Kase's Kinesio taping Manual. For taping, each patient's leg was placed in a relaxed position while he sat on a taping table. The skin was to be free of oils and lotions, to avoid anything that might limit the acrylic adhesive's ability to adhere to the skin. So, the subject's skin was cleaned with alcohol prior to tape application. For the Tibialis anterior, tape was measured from the muscle origin to the insertion while the muscle was stretched. The base of the tape was applied to the origin at the lateral condyle and superior 2/3 of anterolateral surface of tibia. Then the subject was asked to stretch the foot into plantar flexion and eversion; taping was then finished toward the insertion at the medial and plantar surface of medial cuneiform and base of the first metatarsal.
  Arms: Traditional balance exercise + Resistance exercise + Kineso tape

SUMMARY:
The purpose of the study was to compare between effect of whole-body vibration and kineso tape on nerve conduction in patients with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
Diabetes is a huge and rapidly growing health problem worldwide. In 2019, International Diabetes Federation ( IDF) estimated that the number of people with diabetes was 463 million and expected to be 578 million by 2030, and 700 million by 2045. Two-thirds of people with diabetes live in urban areas, and one in five people with diabetes is above 65 year.

Diabetic peripheral neuropathy is the most prevalent complication of diabetes mellitus. The prevalence of DPN ranges from 21.3 to 34.5% in type 2 DM (T2DM) and between seven to 34.2% in type 1 DM (T1DM).

The high incidence and prevalence of falls among older people with type 2 diabetes mellitus were identified as poor diabetic control, diabetic peripheral neuropathy (DPN) and balance impairment.

Study performed by Ahmed et al., reported that Kinesio tape and resistive exercise improve the dorsiflexors and functional performance in diabetic polyneuropathy.

A randomized controlled trial showed that WBV showed beneficial effects on pain, balance, and quality of life in patients with painful Diabetic peripheral neuropathy.

But till know no study reported us whole body vibration better than kineso or vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Patients type 2 diabetes with duration at least 10 years.
* Controlled blood glucose level examined via glycated hemoglobin exam (hba1cless than 9 and more than 6.5).
* Age of patient will range from 50 to 60 years.
* Patients had abnormal nerve conduction study.

Exclusion Criteria:

* Patients having ulceration/infection of feet
* Medical/Surgical conditions limiting functional mobility
* Non-ambulatory patients
* Who are not willing to participate?
* Subjects with Type 1 Diabetes mellitus.
* Subjects with Gestational Diabetes.
* Subjects who are seriously ill.
* Lower limb fracture or trauma
* Significant renal hepatic disorder

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Deep peroneal nerve motor conduction velocity | 6 weeks
  It was measured for all participants in both groups before and after treatment, using Neuropack S1 MEB-9004 NIHON KODEN, JAPAN nerve conduction velocity device.
Sural nerve sensory conduction velocity | 6 weeks
  It was measured for all participants in both groups before and after treatment, using Neuropack S1 MEB-9004 NIHON KODEN, JAPAN nerve conduction velocity device.
Berg Balance Scale | 6 weeks
  It was used to measure the balance for all participants in both groups before and after treatment. It is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. The scale takes approximately 10 to 20 minutes to complete requiring minimal equipment (chair, stopwatch, ruler, and step) and minimal space Berg balance have high validity and reliability. Interpretation: 41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk.
Unilateral Stance Test (UST) | 6 weeks
  It was used to assess postural balance for all participants in both groups before and after treatment. Each subject was instructed to maintain balance on the nondominant leg with eyes opened, eyes closed, and arms spread for as long as possible. The time taken for the contralateral foot to touch the ground was measured in seconds using a stopwatch. This test was performed twice, and the highest score was recorded.
Smartphone Kinesis Balance™ fall prevention app | 6 weeks
  It was used to assess balance and falls risk for all participants in both groups before and after treatment. The app is freely available on the Google Play store, with participants consenting to use of their anonymized data for research and product improvement. The app uses a questionnaire on clinical falls risk factors, combined with a standing balance test and machine learning algorithms to assess balance and falls risk. Participants are provided with advice and exercises to stay healthy and help prevent falls, based on their level of risk (as determined by the smartphone based machine learning algorithm). All data were anonymized at source and transmitted via encrypted channel to a web server where they were stored (in line with GDPR and HIPAA data privacy regulations) for subsequent offline analysis. Data were extracted from the database using MySQL workbench 8.0 (Oracle, CA, USA) and analyzed using Matlab v 9.3.0 (Mathworks, Natick, VA, USA).
Quadriceps femoris muscle strength | 6 weeks
  It was assessed for all participants in both groups before and after treatment, using hand held dynamometry. To evaluate quadriceps muscle strength, the patients were positioned in the prone position, lying with the knee flexed to 90 degrees; the dynamometer was fixed proximal to the ankle on the anterior surface of the leg; and the subjects were asked to perform isometric knee extension. Three maximal isometric contractions were recorded, and the average of the three trials was used for analysis.
Tibialis anterior muscle strength | 6 weeks
  It was assessed for all participants in both groups before and after treatment, using hand held dynamometry. To evaluate tibialis anterior strength, patients were asked to lie supine with their ankles at the edge of the plinth. The ankle joints were placed in the neutral position (between dorsiflexion and plantar flexion). The dynamometer was fixed to the dorsal aspect of the foot, and each subject was asked to perform isometric dorsiflexion. Three maximal isometric contractions were recorded, and the average of the three trials was used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Ezzat Obaya, PhD, Study Chair — Cairo University
Locations (1):
- Lamis Samir Ahmed, Cairo, Egypt